CLINICAL TRIAL: NCT02078622
Title: A Prospective Randomized Controlled Trial to Evaluate the Use of Respiratory Therapists (RTs) to Improve Outcomes and Quality of Life in Patients Diagnosed With COPD
Brief Title: Use of Respiratory Therapists (RTs) to Improve Outcomes and Quality of Life in Patients With COPD
Acronym: RTQOL
Status: Completed | Type: Observational
Sponsor: StratiHealth (Industry)
Responsible Party: Sponsor
Other Study IDs: 20140101S; SH20140101S (Other Grant/Funding Number: STRATIHEALTH)
Record Dates: First submitted 2014-03-01; First posted 2014-03-05 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Respiratory Therapist; Case Management; Education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Case Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- COPD, Education and Case Management: Respiratory Therapist Education and Case Management
  Interventions: Other: Respiratory Therapist Education and Case Management

INTERVENTIONS:
Other: Respiratory Therapist Education and Case Management — Respiratory Therapists will conduct home care visits over a period of one-year at two-week intervals

SUMMARY:
Evaluate subjects in an prospective randomized controlled trial in which subjects will be administered scientifically validated questionnaires to determine the effect of the education and case management by Respiratory Therapists (RTs) on improvements in: health outcomes and quality of life as primary endpoints

Utilize: Chronic Respiratory Disease Questionnaire (CRQ)

The secondary endpoints will be: Rate of exacerbation's, Health care utilization (emergency room encounters, hospital admissions)

DETAILED DESCRIPTION:
Evaluate subjects in an prospective randomized controlled trial in which subjects will be screened and administered scientifically validated questionnaires at study entry and during the observation period at specified intervals to determine the effect of the education and case management by Respiratory Therapists (RTs) on improvements in health outcomes and quality of life as primary endpoints, utilizing the Chronic Respiratory Disease Questionnaire (CRQ). The secondary endpoints will be rate of exacerbation's and health care utilization (emergency room encounters, hospital admissions).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Cognitive ability to retain education and training
* Resides in a stable residence or home, apartment
* Managed by primary care physician (family practice)

Exclusion Criteria:

* Lacks cognitive ability to retain education and training
* Not managed by primary care physician (family practice)
* No stable residence or is homeless

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with COPD
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Quality of Life Using Chronic Respiratory Disease Questionnaire | Measure Dyspnea at baseline upon study entry and change from baseline every two weeks up to three months; Numerical, 7-point modified Likert Scale; Total score and subscores on categories; higher scores indicate better health-related quality of life
  Using the CRQ Evaluate Health Outcomes and QOL

SECONDARY OUTCOMES:
Healthcare Utilization | 1 year
  Hospital Admission, Emergency Room Encounters

CONTACTS AND LOCATIONS:
Overall Officials: ISABEL PEREIRA, MD, Principal Investigator — StratiHealth; VERNON R PERTELLE, RRT, Study Director — StratiHealth
Locations (1):
- Isabel Pereira, Md, Carlsbad, California, United States